CLINICAL TRIAL: NCT00741663
Title: Phase 4 Study on the Comparison Between Combined Versus Sequential Diuretic Treatment of Moderate Ascites in Nonazotemic Patients With Cirrhosis
Brief Title: Spironolactone Versus Spironolactone Plus Furosemide (SVSSF)
Acronym: SVSSF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Prof. Paolo Angeli, Dept. of Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 318P
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Cirrhosis; Ascites
Keywords: cirrhosis; ascites; diuretic therapy; potassium canrenoate; furosemide; hyperkalemia; plasma renin activity; nitric oxide; serum sodium concentration; refractory ascites; Nonazotemic patients with cirrhosis and moderate ascites
MeSH Terms: conditions — Fibrosis; Ascites; Hyperkalemia | interventions — Spironolactone; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Spironolactone and furosemide
- B (Experimental)
  Interventions: Drug: Spironolactone and furosemide

INTERVENTIONS:
Drug: Spironolactone and furosemide — Patients in arm A will receive potassium canrenoate at the initial dose of 200 mg/day, then increased up to 400 mg/day. Non responders will be treated with 400 mg/day of potassium canrenoate and furosemide at an initial dose of 50 mg/day, then increased up to 150 mg/day.
  Arms: A
Drug: Spironolactone and furosemide — Patients in arm B will receive at first 200 mg/day of potassium canrenoate and 50 mg/day of furosemide, then increased up to 400 mg/day and 150 mg/day, respectively.

SUMMARY:
The question whether the sequential diuretic therapy, that means using an antialdosteronic drug at first and adding a loop diuretic in nonresponders, is better than the combination of the two diuretics from the beginning (combined diuretic therapy) in the treatment of ascites in patients with cirrhosis is still open. Therefore, the aim of the study is to compare sequential versus combined diuretic therapy in these patients. One hundred patients will be randomized into two groups. Group A will receive potassium canrenoate at the initial dose of 200 mg/day, then increased up to 400 mg/day. Non responders will be treated with 400 mg/day of potassium canrenoate and furosemide at an initial dose of 50 mg/day, then increased up to 150 mg/day. Group B will receive at first 200 mg/day of potassium canrenoate and 50 mg/day of furosemide, then increased up to 400 mg/day and 150 mg/day, respectively.

The percentage of responders to dthe diuretic treatment, the time to get the resolution of ascites and the rate of adverse effects will be compared between the two Groups of Patients.

ELIGIBILITY:
Inclusion Criteria:

* Grade 2 ascites
* Serum creatinine less than 1.2 mtg/dl
* Serum sodium > 130 mmol/l
* Serum potassium within 3.5 and 4.5 mmol/l
* At least five days after the withdrawal of diuretics
* A 90 mmol/day Na diet.

Exclusion Criteria:

* Any therapeutic paracentesis for ascites before inclusion
* Cardiac or respiratory disease
* Gastrointestinal bleeding, hepatic encephalopathy, bacterial infections in the last 4 weeks before inclusion.
* The use of NSAIDs or other nephrotoxic drugs in the last 4 weeks before inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
the percentage of responders to the diuretic treatment; the percentage of patients who develop adverse effects to diuretics | within three weeks
the percentage of patients who will respond to the diuretic treatment, the percentage of patients who will develop adverse effects to diuretics | within three weeks

SECONDARY OUTCOMES:
time to get the response to diuretics | within three weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Padova, Dept. of Clinical and Experimental Medicine, Padua, Italy

REFERENCES:
- [Result] Santos J, Planas R, Pardo A, Durandez R, Cabre E, Morillas RM, Granada ML, Jimenez JA, Quintero E, Gassull MA. Spironolactone alone or in combination with furosemide in the treatment of moderate ascites in nonazotemic cirrhosis. A randomized comparative study of efficacy and safety. J Hepatol. 2003 Aug;39(2):187-92. doi: 10.1016/s0168-8278(03)00188-0. PMID 12873814
- [Derived] Angeli P, Fasolato S, Mazza E, Okolicsanyi L, Maresio G, Velo E, Galioto A, Salinas F, D'Aquino M, Sticca A, Gatta A. Combined versus sequential diuretic treatment of ascites in non-azotaemic patients with cirrhosis: results of an open randomised clinical trial. Gut. 2010 Jan;59(1):98-104. doi: 10.1136/gut.2008.176495. PMID 19570764